CLINICAL TRIAL: NCT05692999
Title: Maintenance Pembrolizumab at Usual or Low doSE in Non-squamous Lung Cancer: a Non-inferiority Study
Acronym: Pulse
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-006795-16; 2021/3336 (Other: CSET number); 2023-503481-23-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-20; First posted 2023-01-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non-squamous Lung Cancer
MeSH Terms: interventions — pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse Arm (Experimental)
  Interventions: Drug: Pembrolizumab 200 mg Q6W; Drug: Pemetrexed 500 mg/m^2 Q3W
- Control Arm (Active Comparator)
  Interventions: Drug: Pemetrexed 500 mg/m^2 Q3W; Drug: Pembrolizumab 200 mg Q3W or 400 mg Q6W

INTERVENTIONS:
Drug: Pembrolizumab 200 mg Q6W — Pembrolizumab 200mg Q6W
  Arms: Pulse Arm
Drug: Pemetrexed 500 mg/m^2 Q3W — Pemetrexed 500 mg/m^2 Q3W
Drug: Pembrolizumab 200 mg Q3W or 400 mg Q6W — Pembrolizumab 200 mg Q3W or 400 mg Q6W
  Arms: Control Arm

SUMMARY:
Pulse is a randomized non-inferiority phase III clinical trial assessing a new mode of immunotherapy administration based on increased interval time between 2 infusions as maintenance treatment in Pulse arm compared with the conventional administration in Control arm.

In both treatment arms, pembrolizumab alone or combined with pemetrexed is allowed as maintenance treatment. Indeed :

In Pulse arm : Pembrolizumab 200 mg will be administered to patients every 6 weeks (Q6W) plus, in the absence of contra-indication pemetrexed 500 mg/m^2 will be administered every 3 weeks (Q3W).

In control arm : Pembrolizumab 200 mg will be administered to patients every 3 weeks (Q3W) or 400 mg every 6 weeks plus,in the absence of contra-indication pemetrexed 500 mg/m^2 will be administered every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria:

A) To be checked before the induction phase (only for patient included before induction phase) :

1. Histologically or cytologically confirmed diagnosis of non-squamous non-small cell lung cancer (NSCLC).
2. Non-operable / non-irradiable stage III or stage IV.
3. Patient must be eligible to receive 3 or 4 cycles of induction treatment combination with pembrolizumab plus platinum (cisplatin or carboplatin) and pemetrexed.
4. In the presence of an EGFR mutation, an ALK or ROS1 rearrangement the patient must have received at least one specific targeted therapy line.
5. Age ≥ 18 years old.
6. Performance status 0 or 1.
7. Signed informed consent.
8. Patient affiliated to a social security system or beneficiary of the same.

B) To be checked before the maintenance phase (for all patient) :

1. Histologically or cytologically confirmed diagnosis of non-squamous non-small cell lung cancer (NSCLC).
2. Non-operable / non-irradiable stage III or stage IV.
3. Received 3 or 4 cycles of induction treatment combination with pembrolizumab plus platinum (cisplatin or carboplatin) and pemetrexed.
4. Patient must be eligible to receive maintenance pembrolizumab with or without pemetrexed, last induction chemotherapy cycle within 42 days before randomization.
5. Stable disease, partial or complete response according to RECIST 1.1 criteria after induction chemotherapy and pembrolizumab. Targets lesions are not required before randomization.
6. In the presence of an EGFR mutation, an ALK or ROS1 rearrangement the patient must have received at least one specific targeted therapy line (not needed a second time if already checked before induction phase).
7. Patients with baseline brain metastases will be eligible in case of stability or no evidence of progression and if they remain clinically stable.
8. Age ≥ 18 years old.
9. Performance status 0 or 1.
10. Signed informed consent (only for patient included after induction phase).
11. Patient affiliated to a social security system or beneficiary of the same.
12. Creatinine clearance > 30 ml/min by Cockcroft-Gault* or MDRD in case that patient will start maintenance just with pembrolizumab but ≥ 45 ml/min if the patient will receive pemetrexed plus pembrolizumab.

    *Cockcroft- Gault Formula:
    * Female CrCl = [(140 - age in years) x weight in kg x 0.85] / 72 x serum creatinine in mg/dL;
    * Male CrCl = [(140 - age in years) x weight in kg x 1.00] /72 x serum creatinine in mg/dL.
13. Neutrophils ≥ 1500/μL and platelets ≥ 100 000/μL.
14. Bilirubin ≤ 1.5 upper limit normal (ULN).
15. Transaminases, Alkaline phosphatase ≤ 2.5 x the ULN except in case of liver metastases (5 x ULN).
16. Patients might have received platinum-based chemotherapy as an adjuvant or neoadjuvant treatment, or with radiotherapy for a localized lung cancer, provided that the chemotherapy was ended more than 6 months before the first cycle of induction chemotherapy.
17. Patients might have received previous immune checkpoint inhibitors as an adjuvant or neoadjuvant treatment, or as a consolidation treatment after radiotherapy for a localized lung cancer, but the immune checkpoint inhibitors must be finished at least than 12 months before the first cycle of induction chemotherapy for advanced stage.
18. A woman is eligible for the study if she is no longer likely to procreate (physiologically unfit to carry out a pregnancy), which includes women who have had: a hysterectomy, an oophorectomy, a bilateral tubal ligation.

    Post-menopausal women:
    * Patients not using hormone replacement therapy should have had a complete cessation of menstruation for at least one year and be over 40 years of age, or, if in doubt, have an FSH (Follicle Stimulating Hormone) level > 40 mIU/mL and an estradiol level < 40 pg/mL (< 150 pmol/L).
    * Patients using hormone replacement therapy must have had a complete cessation of menstruation for at least one year and be over 45 years of age or have evidence of menopause (FSH and estradiol levels) before starting hormone replacement therapy.
19. Women who are likely to procreate are eligible if they have a negative serum pregnancy test in the week before the first dose of treatment and preferably as close as possible to the first dose and if they agree to use an effective contraceptive method during the course of the study through 4 months after the last dose of study medication.

Sexually active males patients must agree to use condom during the study and for at least 4 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.

Exclusion Criteria:

A) To be checked before the induction phase (only for patient included before induction phase) :

1. Mixed small-cell, squamous-cell carcinoma.
2. Mental or psychological illness that does not allow the patient to give informed consent.
3. Pregnant or breastfeeding women.
4. History of HIV or chronic hepatitis B or C.
5. Active or uncontrolled infection.
6. History of one or more of the following cardiovascular disorders in the previous 6 months:

   * Coronary artery bypass or peripheral arterial bypass, cardiac angioplasty or stent.
   * Myocardial infarction
   * Severe or unstable angina pectoris
   * Peripheral vascular disease, pulmonary embolism or untreated thromboembolic events, stroke or transient ischemic attack. Note: Patients with recent deep vein thrombosis (including pulmonary embolism) treated with anticoagulant for at least 4 weeks and clinically stable are eligible.
   * Congestive heart failure class III or IV as defined by the NYHA
7. Concomitant treatment with another experimental treatment or participation in another clinical trial.

B) To be checked before the maintenance phase (for all patient) :

1. Presence of grade 3 or 4 toxicity related to pembrolizumab limiting maintenance treatment continuation.
2. Mixed small-cell, squamous-cell carcinoma.
3. Corticosteroids at a dose greater than 20 mg per day of prednisone or equivalent.
4. Patient unable to follow the therapeutic program.
5. Mental or psychological illness that does not allow the patient to give informed consent.
6. Pregnant or breastfeeding women.
7. Ongoing immunosuppressive systemic therapy (cyclophosphamide, aziatropin, methotrexate, thalidomide and anti-TNF).
8. Active autoimmune diseases. History of autoimmune diseases including myasthenia gravis, lupus erythematosus, rheumatoid arthritis, irritable bowel syndrome, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis. Patients with a history of autoimmune hypothyroidism treated with a stable dose of hormone replacement therapy are eligible. Patients with diabetes treated with insulin are eligible.
9. History of idiopathic pulmonary fibrosis, organized pneumonia (i.e., obliterating bronchiolitis), drug-induced lung disease or active signs of pneumonia, pulmonary infiltration (regardless of cause) detected on the baseline chest CT-scan.
10. History of any other hematologic or primary solid tumor malignancy unless in remission for at least 2 years and without specific treatment (as example, not allowed hormonal therapy to replace for breast cancer or hormonal therapy substitution in prostate cancer). pT1-2 prostatic cancer Gleason score < 6, superficial bladder cancer, non-melanoma skin cancer or carcinoma in situ of the cervix are allowed.
11. Presence of a condition or condition that makes patient participation in the study inappropriate, including serious unresolved or unstable toxicities from previous administration of another experimental treatment or any medical condition that could interfere with patient safety, obtaining consent or compliance with study procedures.
12. Administration of a live attenuated vaccine within the 4 weeks before day 1 of Cycle 1 or administration of a live attenuated vaccine planned for the duration of the study. The flu vaccine can be given during the flu season (approximately from October to May). Patients should not receive a live attenuated influenza vaccine during the 4 weeks preceding day 1 of Cycle 1 and should not receive this type of vaccine during the study.
13. History of HIV or chronic hepatitis B or C (not needed a second time if already checked before induction phase).
14. Active or uncontrolled infection.
15. History of one or more of the following cardiovascular disorders in the previous 6 months:

    * Coronary artery bypass or peripheral arterial bypass, cardiac angioplasty or stent.
    * Myocardial infarction
    * Severe or unstable angina pectoris
    * Peripheral vascular disease, pulmonary embolism or untreated thromboembolic events, stroke or transient ischemic attack. Note: Patients with recent deep vein thrombosis (including pulmonary embolism) treated with anticoagulant for at least 4 weeks and clinically stable are eligible.
    * Congestive heart failure class III or IV as defined by the NYHA
16. Concomitant treatment with another experimental treatment or participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1166 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 years
  defined as the time elapsed between the date of randomization and the date of death whatever the cause. Patients alive at the date of last follow-up will be censored at that date.

SECONDARY OUTCOMES:
Progression-free survival | 6 years
  defined by the time between the randomization date and the date of observation of a progression of the disease according to RECIST 1.1 or death of the patient (all causes combined) or date of last follow-up if the patient is alive without progression or lost to follow up.
Duration of response between both treatment arms. | 6 years
  Duration of response among patients who had a response (CR/PR) after the 4 induction cycles. It is defined by the time between first response observed (i.e. randomization date) and first event observed (progression, secondary malignancy or death in case of no previous progression).
Assessment of quality of life between both treatment arms via the EORTC QLQ-C30 questionnaire. | 6 years
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life questionnaire (EORTC QLQ-C30).
  The EORTC QLQ-C30 was developed to assess the quality of life of cancer subjects and is the most widely used cancer-specific HRQoL instrument. It contains 30 items and measures five functional dimensions (physical, role, emotional, cognitive, and social), three symptom items (fatigue, nausea/vomiting, and pain), six single items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact) and global health and quality of life. The global health and quality of life scale uses a 7-point scale scoring with anchors (1=very poor and 7=excellent); the other items are scored on a 4 point scale (1=not at all, 2=a little, 3= quite a bit, 4=very much).
Assessment of quality of life between both treatment arms via the EORTC QLQ-LC13 questionnaire. | 6 years
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC13).
  The EORTC QLQ-LC13 covers 13 typical symptoms of lung cancer patients, such as coughing, pain, dyspnea, sore mouth, peripheral neuropathy, and hair loss. It is scored on a 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much).
Assessment of quality of life between both treatment arms via the EQ-5D-5L questionnaire. | 6 years
  Patient reported outcomes via the 5-level EuroQol-5D (EQ-5D-5L questionnaire).
  The EQ-5D-5L essentially consists of five health state dimensions include the following: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-point scale from 1 (extreme problem) to 5 (no problem). The EQ-5D-5L also includes a graded (0 = The worst health you can imagine, to 100 = The best health you can imagine) vertical visual analog scale on which the subject rates his or her general state of health at the time of the assessment.
Treatment tolerance in both treatment arms | 6 years
  Frequency of adverse events according to CTCAE V5
Economic evaluation | 6 years
  An important cost reduction per patient associated to treatment de-escalation is expected. We will compare the costs between the two arms. Time horizon extends from randomization to the date of last follow-up.
  Direct medical costs will be estimated from the French national health insurance perspective (Système National des Données de Santé, SNDS).
Population pharmacokinetic analysis in both arms (primary objective) | 6 years
  The primary objective of the PK study will be to evaluate the systemic exposition (Ctrough) of pembrolizumab in both arms.
Population pharmacokinetic analysis in both arms (secondary objective) | 6 years
  The secondary objective of the PK study will be to use the clearance evolution of the pembrolizumab as marker of the response to explore the potential correlation between clearance evolution and the survival.
Evaluate the saturation of PD-1 on circulating lymphocytes in both arms | 6 years
  Calculate the % of saturation of PD-1 on fresh circulating lymphocytes at baseline and during treatment in both arms.
Evaluate the target engagement pharmacodynamics (PD) in both arms | 6 years
  Target engagement pharmacodynamics (PD) will be assayed using the interleukin-2 (IL-2) stimulation ratio at baseline and during treatment in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BESSE, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (37):
- CHU UCL Namur - Site Sainte Elisabeth, Namur, Belgium
- France (30):
  - Centre Hospitalier de Carcassonne, Carcassonne, Aude
  - Clinique Sainte Anne - Strasbourg, Strasbourg, Bas-Rhin
  - Institut de Cancérologie Strasbourg Europe (ICANS), Strasbourg, Bas-Rhin
  - Hôpital Européen de Marseille, Marseille, Bouches-du-Rhône
  - Groupe Hospitalier La Rochelle, La Rochelle, Charente-Maritime
  - Centre Hospitalier Régional Universitaire de Brest (Hôpital Morvan), Brest, Finistère
  - Centre Hospitalier des Pays de Morlaix, Morlaix, Finistère
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace, Mulhouse, Haut-Rhin
  - Centre Hospitalier de Bigorre, Tarbes, Hautes-Pyrénées
  - Hôpital Foch, Suresnes, Hauts-de-Seine
  - Centre Hospitalier de Béziers, Béziers, Hérault
  - CHU Rennes, Rennes, Ille-et-Vilaine
  - Centre Hospitalier de Saint-Malo, St-Malo, Ille-et-Vilaine
  - Centre Hospitalier Régional Universitaire de Tours, Tours, Indre-et-Loire
  - Centre Hospitalier Universitaire - La Réunion - Site Felix Guyon, Saint-Denis, La Réunion
  - Centre Hospitalier Universitaire - La Réunion - Site Sud, Saint-Pierre, La Réunion
  - Centre Hospitalier Régional d'Orléans - NHO, Orléans, Loiret
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron, Lyon
  - Centre Hospitalier de Cholet, Cholet, Maine-et-Loire
  - Centre Hospitalier Intercommunal de Compiègne-Noyon, Compiègne, Oise
  - CHU St-Etienne, Saint Priest En Jarez, Pays de la Loire Region
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrénées-Atlantiques
  - Centre Hospitalier Intercommunal Créteil, Créteil, Val-de-Marne
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé, Val-de-Marne
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - Centre Hospitalier d'Auxerre, Auxerre, Yonne
  - Hôpital Pitié-Salpêtrière - APHP, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital Tenon - APHP, Paris
  - Hôpital Paris Saint-Joseph, Paris
- Spain (6):
  - H. Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - H. Clinico San Carlos, Madrid
  - HU. 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - H.Virgen del Rocio, Seville